CLINICAL TRIAL: NCT01549132
Title: Non-invasive Retinal Oximetry Using Oxymap in Patients With Diabetic Maculopathy Receiving Laser/Intravitreal Anti-VEGF Therapy
Brief Title: Retinal Oximtery Following Treatment for Diabetic Maculopathy
Status: Completed | Type: Observational
Sponsor: East Kent Hospitals University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: EKHT RETINAL RESEARCH UNIT
Record Dates: First submitted 2012-03-06; First posted 2012-03-09 (Estimated); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Diabetic Maculopathy
Keywords: Clinically significant macular oedema; Retinal Oximetry; Spectral imaging; Retinal Laser therapy; Intravitreal Anti-VEGF Injection therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators believe that oxygen saturation measurements in the retina may provide more information on how well the retina is working and may detect problems in the retina earlier than the fundus fluorescein angiography (FFA). This may be useful to an ophthalmologist so that they may identify abnormal areas of the retina and commence or change the treatment so that they may prevent irreversible blindness.

Most patients with clinically significant macular oedema and/or ischaemic diabetic retinopathy could have either laser or Intravitreal Anti-VEGF injection treatment provided they are counseled about the risks. It is known the Anti-VEGF injections reduce oedema and it is believed that laser treatment of the retina in this condition improves the oxygen supply to the retina and sometimes reverses the damage. It will be useful to take pictures of these treated eyes using the Oxymap spectral retinal camera(s) to see whether the investigators can detect a change in the oxygen saturation in the retina before and after treatment using our oxygen saturation methods.

DETAILED DESCRIPTION:
WHAT IS SPECTRAL IMAGING?

This is a way of studying in detail an area that is being imaged. This can be done because each picture of the same area is taken using different colours of light (wavelength). Different materials in the picture will absorb and reflect the different wavelengths of light from a hyperspectral camera differently. It is then possible to look at each point in the picture and work out what is in the picture. This has been used in satellites and aeroplanes to identify what is on the ground. For example, it can distinguish the different types of trees on the ground based on the different way they absorb and reflect different wavelengths of light.

USING SPECTRAL IMAGING IN MEDICINE. Spectral imaging was found to have uses in medicine because of its ability to distinguish one thing from another. A lot of Spectral imaging research has been done to measure the amount of oxygen in the blood. This is because oxygen is important to all living cells in the human body - without it cells would die or stop working. Oxygen is carried to living cells by blood in blood vessels known as arteries and the left over is carried away by veins. Most of the oxygen in the blood is transported by cells in the blood containing a chemical called haemoglobin. There are two main forms of haemoglobin called oxyhaemoglobin (haemoglobin binds to oxygen) and deoxyhaemoglobin (haemoglobin that is not bound to oxygen). The proportion of oxyhaemoglobin to the total amount of haemoglobin (both oxyhaemoglobin and deoxyhaemoglobin) is called the oxygen saturation and is presented as a percentage. The normal saturation in the artery is about 97% because it contains more oxyhaemoglobin and in the vein it is about 75% because it contains less oxyhaemoglobin. Importantly oxyhaemoglobin (HbO2) and deoxyhaemoglobin (Hb) have different spectral characteristics - i.e they absorb light differently at various wavelengths of light. This has been extensively documented in various publications using samples of blood. This property is the basis of pulse oximetry which is the measurement of the oxygen saturation (OS) in the finger tip using a saturation probe which is commonly used in the hospital.

The different spectral characteristics of Hb and HbO2 can also be used in spectral imaging to calculate the amount of each in the blood to perform oxygen saturation measurements in certain parts of the body. This has previously been used to study the oxygen supply in the skin and also to look at the oxygen supply in patients with diabetes which is a condition that is caused by a lack of a hormone called insulin causing high amount of sugar in the blood resulting in damage to the blood vessels.

Spectral imaging has only recently started to be used in imaging the eye. The main emphasis of Spectral imaging in ophthalmology has been on measuring the oxygen saturations in the retina (the layer at the back of the eye that allows us to see). This is called retinal oximetry. In essence, the principles of retinal oximetry are similar to that of pulse oximetry, i.e using the different spectral characteristics of Hb and HbO2 to calculate the oxygen saturation.

In diabetic retinopathy, the only way the investigators can study the blood supply is by performing a Fundus Fluorescein Angiogram (FFA). This is an invasive test which involves the injection of a dye into the arm, this dye is transported by blood to the eye and pictures of the blood vessels are taken with the dye in it. Also, importantly, there are side effects (sometimes life-threatening) to injecting this dye into the arm. If there is a problem with the blood supply in the retina then the dye will not fill up in the blood vessel and is seen in the pictures as a black area. The FFA provides information on the blood supply but not directly on the amount of oxygen in it. Loss of sight from diabetic retinopathy and age-related macular degeneration is believed to be caused by a reduction in the amount oxygen being supplied to the retina by the blood vessels.

The investigators believe that oxygen saturation measurements in the retina using spectral imaging could be a more useful test for an ophthalmologist because it may provide more information on how well the retina is working and may detect problems in the retina earlier than the FFA. This may be useful to an ophthalmologist so that they may identify abnormal areas of the retina and commence or change the treatment so that they may prevent irreversible blindness.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic Retinopathy affecting the central retina (designated maculopathy)
* No contraindications to pupil dilation
* Ocular media sufficiently clear to enable retinal imaging
* Pupils which can be dilated (i.e not using miotic medication)
* Willingness to participate with the research study and formal consent obtained.

Exclusion Criteria:

* Narrow drainage angles or any other contraindication to being dilated.
* Dense cataracts or other ocular media opacities inhibiting a good view of the retina on fundoscopy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: • Patients will be selected from the Ophthalmology clinics with all sites at East Kent Hospitals University Foundation NHS Trust. These patients will be selected non-randomly by the ophthalmology clinician involved in their care based whether their clinical diagnosis fulfils the inclusion criteria. The ophthalmologists who are seeing patients in the ophthalmology clinics will identify the patients fulfilling the inclusion criteria for this study.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2012-04; Primary Completion 2013-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Retinal oximetry differences in patients with sight threatening diabetic macular oedema after treatment | 1 year
  Does retinal oxygen levels in small blood vessels as measured by spectral imaging photography using the oxymap device at the centre of the retina (macula) differ in diabetic retinopathy in sight threatening disease?

CONTACTS AND LOCATIONS:
Overall Officials: NISHAL PATEL, MD FRCOPHTH, Principal Investigator — CONSULTANT OPHTHALMOLOGIST